CLINICAL TRIAL: NCT07244718
Title: Effects of Music-Assisted Progressive Muscle Relaxation on Sleep Quality, Fatigue, Emotional Symptoms, and Quality of Life in Sedentary Obese Women
Brief Title: Investigation of The Effect of Progressive Muscle Relaxation Technique in Sedentary Obese Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Raziye Şavkın, Assoc. Prof., Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-60116787-020-481634
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Progressive Muscle Relaxation Technique
Keywords: Progressive Muscle Relaxation Technique; Sleep Quality; Mood; Fatique; Quality of Life; Obesity
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Other): Participants in the control group will not receive any therapeutic intervention during the study period. To equalize the time and attention provided to the intervention group, participants will be instructed to lie down in a comfortable position for twenty to thirty minutes once a day, before going to bed, for a total of six weeks, without performing any relaxation technique or physical activity.
  They will be asked to record each daily session in an activity log and will be instructed not to miss more than two sessions per week. Participants will also be asked to refrain from receiving any additional complementary or mind-body therapies that promote relaxation-such as acupuncture, massage, meditation, or other similar practices-throughout the study period. No restrictions will be placed on their usual daily routines or lifestyle habits.
  After completion of all assessments at the end of the study, participants in the control group will be provided with information about progressive m
  Interventions: Other: Control
- Intervention group (Experimental): At the beginning of the study, participants will be verbally informed about the progressive muscle relaxation technique, its method of application, and associated breathing techniques. Following this introductory session, twenty- to thirty-minute video and audio recordings prepared by the Turkish Psychologists Association, featuring music-assisted progressive muscle relaxation exercises, will be delivered to participants via a smartphone application.
  Participants will be instructed to follow the video and audio recordings once a day, before going to bed, for a period of six weeks. A follow-up meeting will be scheduled two weeks after the initial session to monitor participant compliance, answer questions, and reinforce proper technique.
  Participants will be asked to record each session in an activity log and will be instructed not to skip more than two sessions per week. In addition, they will be asked to refrain from receiving any complementary or relaxation-based therapies, such a
  Interventions: Other: Music-Assisted Progressive Muscle Relaxation

INTERVENTIONS:
Other: Control — No therapeutic intervention will be performed on participants in the control group after baseline assessment. To equalize the time and attention provided to the intervention group, participants in the control group will be asked to lie down in a comfortable position for twenty to thirty minutes once a day before going to bed for six weeks, without engaging in any relaxation technique or physical activity. They will be instructed to record these daily sessions in an activity log and will be asked not to miss more than two sessions per week.
  Participants will also be asked to refrain from receiving any additional complementary therapies that promote relaxation-such as acupuncture, massage, and other mind-body techniques-throughout the study period. No restrictions will be placed on their usual daily routines or lifestyle habits.
  After completion of all study assessments, participants in the control group will be informed about progressive muscle relaxation techniques, including their a
  Arms: Control group
Other: Music-Assisted Progressive Muscle Relaxation — At the beginning of the study, participants will be verbally informed about the progressive muscle relaxation technique, its application steps, and associated breathing techniques. Following this introduction, twenty- to thirty-minute video and audio recordings prepared by the Turkish Psychologists Association-featuring music-assisted progressive muscle relaxation instructions-will be sent to participants via a smartphone application.
  Participants will be instructed to follow the video/audio recordings once a day, before going to bed, for a period of six weeks. Approximately two weeks after the initial meeting, a follow-up session will be scheduled to assess participants' adherence to the protocol and to address any questions or difficulties they may have.
  Throughout the intervention period, participants will be asked to document each session in an activity log and will be instructed not to skip more than two sessions per week. They will also be asked to refrain from receiving any ad
  Arms: Intervention group

SUMMARY:
Obesity is a major public health problem that reduces quality of life and increases the risk of many chronic diseases. Its global prevalence continues to rise, and it is estimated that approximately 18 percent of men and 21 percent of women will be affected by the year 2025. The development and progression of obesity are influenced by individual characteristics such as age, lifestyle, and gender. Women experience hormonally driven changes in body fat across different life stages, including puberty, reproductive years, and the postpartum period, which place them at higher metabolic risk.

Progressive muscle relaxation, particularly when combined with music, has been shown to reduce sleep problems, emotional disturbances, fatigue, and limitations in quality of life across different clinical populations. However, the effectiveness of music-assisted progressive muscle relaxation in sedentary obese women has not been clearly demonstrated.

This study investigates whether a six-week, home-based music-assisted progressive muscle relaxation program can improve sleep quality, emotional well-being, fatigue, and health-related quality of life in sedentary obese women. The intervention can be performed independently in the participants' own living environment, which supports sustainability and enhances self-management. Demonstrating the effectiveness of this method may offer healthcare professionals a low-cost, accessible, non-pharmacological treatment option to improve both physical and emotional well-being in this high-risk population.

ELIGIBILITY:
Inclusion Criteria:

* Female participants aged 18-50 years
* Classified as sedentary according to the International Physical Activity Questionnaire-Short Form (IPAQ-SF)
* Obese, defined as BMI ≥ 30 kg/m²
* Ability to understand written and spoken Turkish
* Ability to comprehend study instructions
* Active use of WhatsApp or Telegram to receive intervention materials

Exclusion Criteria:

* Cognitive impairment affecting communication
* Pregnancy, postpartum period, or lactation
* Use of weight-loss medications or sedative-hypnotic drugs
* Not having a regular menstruation cycle
* Hearing impairment

Criteria for Withdrawal:

* Voluntary withdrawal from the study
* Development of a condition preventing continuation of participation
* Failure to attend sessions regularly (missing more than two sessions per week)
* Incomplete final assessments

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 20 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index | Baseline (Week 0) and Week 6
  The scale designed to assess sleep quality consists of a total of 24 questions. Nineteen of these questions are answered by the individual, while five are answered by their spouse or roommate. The last five questions are not included in the scoring. The total scale score, ranging from 0 to 21, is obtained by summing the scores of seven subcomponents classified as subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, sleep medication use, and daytime dysfunction. A total score of ≤5 indicates good sleep quality, while a score >5 indicates impaired sleep quality.
Nottingham Health Profile | Baseline (Week 0) and Week 6
  The Nottingham Health Profile aims to assess quality of life. It is divided into two sections. The first section consists of six sub-dimensions and 38 items: pain, emotional reactions, sleep, social isolation, physical activity, and energy level. Each sub-dimension score ranges from 0 to 100, and the total score for the first section ranges from 0 to 600. The second section consists of seven items containing questions about areas of life affected by health status. The total score for the second section ranges from 0 to 7. In the evaluation of the scale, low scores are interpreted as minimal impact from the disease, while high scores indicate significant impact.
Chalder Fatigue Scale | Baseline (Week 0) and Week 6
  The Chalder Fatigue Scale assesses the fatigue experienced by individuals over the past month. It consists of 11 items. A high total score on the scale indicates a high level of fatigue.
Depression Anxiety Stress Scale-21 | Baseline (Week 0) and Week 6
  The Depression Anxiety Stress-21 Scale is a shortened version of the Depression Anxiety Stress-42 Scale. It consists of seven items measuring depression, stress, and anxiety. The scale cannot be expressed as a single score; the scores from the three subscales are evaluated separately.
Epworth Sleepiness Scale | Baseline (Week 0) and Week 6
  It was developed to assess the general level of daytime sleepiness during different daily activities. The scale consists of 8 items scored from 0 to 3. The scale score ranges from 0 to 24. The total score of the scale is positively correlated with the person's daytime sleepiness.

OTHER OUTCOMES:
Fatigue Severity Scale | Baseline (Week 0) and Week 6
  The scale contains nine items scored from 1 (strongly disagree) to 7 (strongly agree). The total score is calculated as the mean of all items. Scores <4 indicate absence of fatigue, whereas scores ≥4 indicate clinically relevant fatigue; higher values denote greater fatigue severity.

CONTACTS AND LOCATIONS:
Overall Officials: Raziye ŞAVKIN, Assoc. Prof., Study Chair — Pamukkale University; Beyza Hilal TOY, Msc. PT., Principal Investigator — Pamukkale University; Ummuhan BAŞ ASLAN, Prof., Principal Investigator — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No